CLINICAL TRIAL: NCT05980728
Title: The Prognostic Value of Biomarker in Connective Tissue Disease Patients With Pulmonary Hypertension
Brief Title: Connective Tissue Disease Patients With Pulmonary Hypertension
Status: Not yet recruiting | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: JSPH cohort
Record Dates: First submitted 2023-07-03; First posted 2023-08-08 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Connective Tissue Diseases; Pulmonary Hypertension
Keywords: prognosis , biomarker, pulmonary hypertension
MeSH Terms: conditions — Connective Tissue Diseases; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — DNA RNA Peripheral blood mononuclear cells, Serum, Plasma, Urine,Stool
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Connective Tissue Disease Patients With Pulmonary Hypertension: Connective Tissue Disease Patients With Pulmonary Hypertension
  Interventions: Other: No Intervention
- Connective Tissue Disease Patients Without Pulmonary Hypertension: Connective Tissue Disease Patients Without Pulmonary Hypertension
  Interventions: Other: No Intervention
- healthy: healthy people
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
Adult patients with suspected or confirmed Connective Tissue Disease Patients (CTD)With Pulmonary Hypertension(PH)will be recruited. Patients will be approached, consented, have baseline demographics, diagnostics and disease activity measures recorded, and blood taken. The collection of data and biological material will mirror usual clinical practice as far as possible. Subjects will ideally attend further visits at 3, 6 and 12 months to have bloods taken, outcome measures recorded and questionnaires completed.

ELIGIBILITY:
Inclusion Criteria:

* Definite diagnosis of CTD included Systemic lupus erythematosus（SLE） diagnosed according to the 2019 The European Alliance of Associations for Rheumatology（EULAR） criteria, primary Sjogren's syndrome (pSS) defined according to the 2016 American College of Rheumatology(ACR) criteria, Systemic Sclerosis(SSc) defined according to the 2013 ACR criteria, mixed connective tissue disease (MCTD) defined by Sharp criteria, and Rheumatoid Arthritis(RA) defined according 2010 ACR criteria of two or more CTD at the same time were defined as having overlap syndrome (OS). Patients who had clinical and serological manifestations suggestive of systemic autoimmune diseases but did not fulfil the classification criteria for CTD were defined as having undifferentiated CTD (UCTD).
* PAH was diagnosed by right heart catheterization was defined as mean Pulmonary Artery Pressure (mPAP)>20 Millimeters of mercury（mmHg）, Pulmonary Artery Wedge Pressure（PAWP）≤15mmHg, Pulmonary Vascular Resistance（PVR）>2 Wood

Exclusion Criteria:

* significant interstitial lung disease or chronic obstructive pulmonary disease;
* left heart disease or congenital heart disease associated with pulmonary hypertension;
* chronic thromboembolic pulmonary hypertension;
* portal hypertension;
* drug or toxin exposure;
* HIV infection;
* any other diseases known to be associated with PAH;
* age<18 years.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Connective Tissue Disease Patients With Pulmonary Hypertension
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Death | 30 years
  number of participants with All cause death

SECONDARY OUTCOMES:
Clinical worsening | 30 years
  number of participants with Hospitalization for worsening pulmonary arterial hypertension(PAH),lung or heart/lung transplant) or unsatisfactory long-term clinical response (the 6-minute walk distance decreased > 15% from baseline and World Health Organization(WHO) functional class III/IV symptoms assessed at two clinic visits separated by > 6 months after sufficient PAH targeted drug treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Wang, MD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dai J, Ma L, Zhang Y, Shan L, Li D, Li L, Hu Q, Zhou Z, Sun X, Wang Q, Zhou L. The prognostic value of HFA-PEFF score in connective tissue disease-associated PAH: evidence from a cohort study. BMC Cardiovasc Disord. 2025 Apr 5;25(1):258. doi: 10.1186/s12872-025-04691-y. PMID 40188059
- [Derived] Sun X, Zhang Y, Liu T, Zhang H, Zu B, Zhou L, Wang Q, Zhang M. Clinical characteristics of primary SS- and overlap SS-associated pulmonary arterial hypertension: a multicentre retrospective study. Rheumatology (Oxford). 2025 Jun 1;64(6):3618-3625. doi: 10.1093/rheumatology/keaf013. PMID 39792031
- [Derived] Dai J, Liu T, Zhang H, Sun X, Tang Y, Qian W, Zhang Y, Ye H, Shan L, Li L, Du M, Li D, Zhu Y, Ma K, Liu L, Wang Q, Zhou L. Fragmented QRS complex could predict all-cause mortality in patients with connective tissue disease-associated pulmonary arterial hypertension. Rheumatology (Oxford). 2025 Feb 1;64(2):789-797. doi: 10.1093/rheumatology/keae084. PMID 38323656